CLINICAL TRIAL: NCT05083403
Title: A Randomized Trial of the Hypotension Prediction Index in the Cardiac Operating Room and the Intensive Care Unit
Brief Title: HPI (Hypotension Prediction Index) Care Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-19
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-01

CONDITIONS: Cardiopulmonary Bypass Surgery
Keywords: cardiopulmonary bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HPI Arm (Experimental): AcumenTM HPI Software Feature to guide hemodynamic management in cardiac surgery post-CPB
  Interventions: Device: AcumenTM HPI Software Feature
- Non-HPI Arm (Placebo Comparator): Non-protocolized standard of care management per clinician and provider judgement.
  Interventions: Other: Non-protocolized Standard of Care

INTERVENTIONS:
Device: AcumenTM HPI Software Feature — The AcumenTM HPI Feature Software provides the clinician with physiological insight into a patient's likelihood of trending toward a hypotensive event. The AcumenTM HPI Feature Software suite is enabled by the minimally invasive Acumen IQ sensor.
  Arms: HPI Arm
Other: Non-protocolized Standard of Care — Non-protocolized standard of care to treat subjects
  Arms: Non-HPI Arm

SUMMARY:
A prospective single-center randomized controlled trial to determine if guided hemodynamic management with the Acumen HPI technology in the OR and ICU can reduce the mean duration of hypotension in cardiac surgery patients requiring cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are at least 18 years of age
2. Subjects who have signed the Informed Consent Form
3. Subjects with planned pressure monitoring with an arterial line
4. Subjects with planned sternotomy
5. Subjects with planned general anesthesia
6. Subjects who have ASA Physical Status ≤ 4
7. Subjects with planned cerebral oximetry monitoring
8. Subjects with planned overnight hospitalization
9. Subjects with planned cardiopulmonary bypass (CPB) "on-pump" surgery

Exclusion Criteria:

1. Subjects with a physical site area too limited for proper Sensor placement
2. Subjects with contraindications for Arterial Line Placement;
3. Subjects participating in another (interventional) study
4. Subjects in whom an intraoperative MAP target will be < 65 mmHg
5. Subjects with pre-op or pre-pump or post-pump LVEF < 15%
6. Subjects requiring heart transplant
7. Subjects with pre-existing circulatory support devices or planned circulatory support devices post-bypass
8. Subjects requiring emergency surgery
9. Subjects with known or identified severe PAH (defined as pulmonary systolic pressure> 70mmHg or mean pressures > 55mmHg) as determined by a pre-operative echo or intraoperative Swan-Ganz
10. Subjects with cardiovascular instability in the operating room necessitating the need to go back on bypass for a subsequent run

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Assessment if the use of the AcumenTM HPI Feature Software reduces the mean duration of hypotension (defined as MAP < 65mmHg) | From post-bypass period to the first 8-hour ICU period
  Assessment if the use of the AcumenTM HPI Feature Software reduces the mean duration of hypotension (defined as MAP < 65mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No